CLINICAL TRIAL: NCT03224377
Title: Diagnostic Utility of Anti-mutated Citrullinated Vimentin Antibodies,Anti Cyclic Citrullinated Peptide Antibodies and Rheumatoid Factor in Rheumatoid Arthritis
Brief Title: Diagnostic Utility of Anti MCV Antibodies,Anti CCPantibodies and RF in RA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ayat salah, principal investigator, Assiut University
Other Study IDs: ASA
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and serum sampling separated by centrifugation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- rheumatoid arthritis patients: Complete blood count Esr Crp Liver function test Kidney function test Hepatitis markers Rheumatoid factor Urine analysis Anti cyclic citrullinated peptide antibodies Anti mutated citrullinated vimentin antibodies
  Interventions: Diagnostic Test: anti mutated citrullinated vimentin antibodies
- healthy control: Complete blood count Esr Crp Liver function test Kidney function test Hepatitis markers Rheumatoid factor Urine analysis Anti cyclic citrullinated peptide antibodies Anti mutated citrullinated vimentin antibodies
  Interventions: Diagnostic Test: anti mutated citrullinated vimentin antibodies

INTERVENTIONS:
Diagnostic Test: anti mutated citrullinated vimentin antibodies — Blood sampling using ELisa technique
  Other Names: anti cyclic citrullinated peptide antibodies

SUMMARY:
Rheumatoid arthritis (RA) is a chronic systemic disease affecting primarily the synovium, leading to joint damage and bone destruction(Gravallese E,2002). It is probably the most common autoimmune disease, It is three times more common in women compared to men and usually appears in middle age(poulsom and charles, 2016) .Early diagnosis of RA and its early treatment with disease-modifying anti rheumatic drugs lead to better control and less joint damage .therefore,It is very important to find an acceptable serological marker in order to make an early diagnosis and initiate early treatment to avoid complication and disability ( Orozco C,and Olsen,2006)

Various serum biomarkers are used to diagnose RA, including many autoantibodies. However, only rheumatoid factor (RF) and anticyclic citrullinated peptide (anti-CCP) antibodies have wide acceptance (taylor et 2011).

DETAILED DESCRIPTION:
Antibodies targeting citrullinated proteins are found to be highly specific for the diagnosis of RA (Riedmannet al,2005). Citrullinated antigens are thought to play a pivotal role in the pathogenesis of RA as they are expressed in inflamed joints and, anti-citrullinated protein antibodies are present before clinical disease and are highly specific for RA(van Gaalen et al,2005).

These autoantibodies predict clinical and radiological severity and may be implicated in the pathogenesis of RA ;however, they have a high value in the early diagnosis and early treatment of RA ( Agrawal et al ,2007).

Indeed, it has been demonstrated that anti-citrullinated protein antibodies are produced by plasma cells in the synovial tissue, as concentrations are more than seven fold higher in synovial tissue than in serum (Masson et al,2000).

Rheumatoid factor is not specific to RA, as it is present in patients suffering from other autoimmune and infectious diseases, also found in apparently healthy elderly patients(urusm et al, 2008). Anti- CCP has been shown to be a specific prognostic marker for RA and predict the erosive or non-erosive progression of the disease. Overall, anti-CCP antibodies are a useful marker for aiding the diagnosis of early RA, especially in seronegative(RF negative)( poulsom and charles,2007) Thus, it is a useful tool for the optimal therapeutic management of RA patients.

The diagnosis of RA has been improved by the introduction of other standardized immunoassays for the detection of auto-antibodies against different citrullinated antigens as anti-mutated citrullinated vimentin antibodies .Anti-MCV antibodies have been recommended to be better diagnostic marker for early arthritis (Luime et al,2010). Vimentin is an intermediate filament that is widely expressed by mesenchymal cells &Macrophages and easy to detect in the synovium. Modification of the protein occurs in macrophages undergoing apoptosis, and antibodies to citrullinated vimentin may emerge if the apoptotic material inadequately cleared(Khalifa et ai 2013).

A significant correlation has been established between anti-MCV antibodies titers and both the severity of RA and the disease-activity score (DAS28) ,anti-MCV-positive patients exhibited significantly lower reduction in disease activity and a greater number of swollen joints. Thus, it appears that, anti-MCV antibodies may have the advantage of correlating better with disease activity and patient outcome(Al-Shukaili et al,2012)

The anti-mutated citrullinated vimentin antibody ELISA isa recently developed assay for the detection of IgG antibodies to a vimentin-based peptide .Anti-MCV antibody has been reported with a sensitivity of 65-82%, specificity of 80-95%.Anti-MCV antibody concentrations have also been reported as correlating with disease activity score , prognostic for disease severity, and being treatment sensitive, enabling their use in monitoring response to therapy (Bang et al,2006)

ELIGIBILITY:
Inclusion Criteria:

* patients with RA Patients with SLE,Psoriasis and systemic sclerosis as disease control

Exclusion Criteria:

* 1-malignancy patients 2-chronic infection patients as TB and Hepatitis B&C 3_mixed connective tissue diseases

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 80 patient with different rheumatic diseases,40 patients with RA and 20 patients with other rheumatic diseases (disease control),beside 20 healthy subject age and sex matched with the patients as healthy control.
  The patients will be recruited from Internal medicine department and Rheumatology Out patient clinics of Assuit University Hospital .
  All patients will be diagnosed as RA according to 2010 ACR/EULAR rheumatoid arthritis classification criteria.All patients will under go detailed history and compelete examination Generalized muscloskeletal examination and local clinical examination of affected joints e.g number of swollen joints ,number of tender joints,assessment of disease activity and functional disability by 28 joint disease activity score calculator (DAS28).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2017-10-09 (Estimated); Primary Completion 2018-10-09 (Estimated); Study Completion 2019-02-01 (Estimated)

PRIMARY OUTCOMES:
Anti mutated citrullinated vimentin antibodies | at one day of the study
  blood sample using Elisa technique
Anti cyclic citrullinated peptide antibodies | at one day of the study
  blood sample using Elisa technique

SECONDARY OUTCOMES:
rheumatoid factor (RF) antibody | at one day of the study
  blood sampling

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Agrawal S, Misra R, Aggarwal A. Autoantibodies in rheumatoid arthritis: association with severity of disease in established RA. Clin Rheumatol. 2007 Feb;26(2):201-4. doi: 10.1007/s10067-006-0275-5. Epub 2006 Mar 30. PMID 16572283
- [Result] Hayem G, Chazerain P, Combe B, Elias A, Haim T, Nicaise P, Benali K, Eliaou JF, Kahn MF, Sany J, Meyer O. Anti-Sa antibody is an accurate diagnostic and prognostic marker in adult rheumatoid arthritis. J Rheumatol. 1999 Jan;26(1):7-13. PMID 9918234
- [Result] Orozco C, Olsen NJ. Identification of patients with early rheumatoid arthritis: challenges and future directions. Clin Dev Immunol. 2006 Jun-Dec;13(2-4):295-7. doi: 10.1080/17402520600877794. PMID 17162371
- [Result] Poulsom H, Charles PJ. Antibodies to citrullinated vimentin are a specific and sensitive marker for the diagnosis of rheumatoid arthritis. Clin Rev Allergy Immunol. 2008 Feb;34(1):4-10. doi: 10.1007/s12016-007-8016-3. PMID 18270850
- [Result] Riedemann JP, Munoz S, Kavanaugh A. The use of second generation anti-CCP antibody (anti-CCP2) testing in rheumatoid arthritis--a systematic review. Clin Exp Rheumatol. 2005 Sep-Oct;23(5 Suppl 39):S69-76. PMID 16273788
- [Result] Ursum J, Nielen MM, van Schaardenburg D, van der Horst AR, van de Stadt RJ, Dijkmans BA, Hamann D. Antibodies to mutated citrullinated vimentin and disease activity score in early arthritis: a cohort study. Arthritis Res Ther. 2008;10(1):R12. doi: 10.1186/ar2362. Epub 2008 Jan 28. PMID 18226202
- [Result] van Gestel AM, Haagsma CJ, van Riel PL. Validation of rheumatoid arthritis improvement criteria that include simplified joint counts. Arthritis Rheum. 1998 Oct;41(10):1845-50. doi: 10.1002/1529-0131(199810)41:103.0.CO;2-K. PMID 9778226
- [Result] Vossenaar ER, Radstake TR, van der Heijden A, van Mansum MA, Dieteren C, de Rooij DJ, Barrera P, Zendman AJ, van Venrooij WJ. Expression and activity of citrullinating peptidylarginine deiminase enzymes in monocytes and macrophages. Ann Rheum Dis. 2004 Apr;63(4):373-81. doi: 10.1136/ard.2003.012211. PMID 15020330